CLINICAL TRIAL: NCT02247375
Title: A Double-blind, Randomized, Three Parallel Group Placebo-controlled Study to Investigate Pharmacokinetics, Effect on Expression of CD11b/CD18 (Mac-1), as Well as Safety and Efficacy of Two Oral Doses of BIIL 284 BS (Dosage: 25 mg Daily, 150 mg Daily) in Patients With Rheumatoid Arthritis Over Two Weeks
Brief Title: Pharmacokinetics, Safety and Efficacy of BIIL 284 BS in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 543.14
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — amelubant

ARMS (3):
- Low dose of BIIL 284 BS (Experimental)
  Interventions: Drug: Low dose of BIIL 284 BS tablets
- High dose of BIIL 284 BS (Experimental)
  Interventions: Drug: High dose of BIIL 284 BS tablets
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low dose of BIIL 284 BS tablets
  Arms: Low dose of BIIL 284 BS
Drug: High dose of BIIL 284 BS tablets
  Arms: High dose of BIIL 284 BS
Drug: Placebo
  Arms: Placebo

SUMMARY:
Safety, pharmacokinetics, pharmacodynamics [CD11b/CD18 (Mac-1) expression] and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Male and female from 18 to 65 years of age
* Patients suffering from active rheumatoid arthritis as defined by the ARA criteria revised 1987

  --- At least 4 of the following 7 criteria must have been present:
  * morning stiffness in and around the joints lasting at least 1 hour before maximal improvement for at least 6 weeks
  * arthritis (soft tissue thickening or fluid - not bony overgrowth alone) of at least 3 joint areas for at least 6 weeks
  * arthritis of hand joints (at least one area swollen in a wrist, metacarpophalangeal (MCP) or proximal interphalangeal (PIP) joint) for at least 6 weeks
  * symmetric arthritis (observed by a physician) with simultaneous involvement of the joints on both sides of the body for at least 6 weeks
  * rheumatoid nodules (observed by a physician) over bony prominences or extensor surfaces or in juxta-articular regions
  * serum rheumatoid factor positive
  * x-ray changes typical of rheumatoid arthritis (erosions or unequivocal bony decalcification localised in or most marked adjacent to the involved joints)
* Patient belonging to the RA functional class I, II or III
* Patient's written informed consent

Exclusion Criteria:

* Pregnancy (to be excluded by pregnancy test) or breast feeding
* Women of childbearing potential not using adequate contraception
* Treatment with methotrexate in the previous month or intended use during the trial period
* Treatment with slow acting antirheumatic drugs (SAARDs)/disease-modifying antirheumatic drugs (DMARDs) other than parenteral gold, D-penicillamine, sulfasalazine, chloroquine / hydroxychloroquine corticosteroid during the last 2 months prior to study entry
* Treatment with more than one SAARD/DMARD and/or corticosteroid during the last 2 months prior to study entry
* Change in treatment with SAARDs/DMARDs during the last 2 months prior to study entry or intended change during the trial duration
* Change in treatment with corticosteroids during the last month prior to study entry or intended change during the trial duration
* Systemic treatment with corticosteroids at a dose higher than 10 mg/day or 0.2 mg/kg/day (prednisone equivalent), respectively (whichever is lower) during the last month prior to study entry or their intended use during the trial treatment period
* Change in treatment with non-steroidal anti-inflammatory drugs (NSAIDs) during the last month prior to study entry or intended change during the trial duration
* Treatment with EnbrelTM (etanercept) or experimental therapies during the last 3 months prior to study entry
* Synovectomy and/or surgical treatment for RA in the previous month or during the trial
* Clinical evidence of known severe cardiovascular, hepatic, renal, respiratory, metabolic, haematological, immunological, gastro-intestinal, hormonal or mental disorders
* Any other rheumatological or non-rheumatological disease that could interfere with the evaluation of efficacy and safety
* Patients with active malignant disease
* Patients with chronic or acute infections during the previous month
* Patients with abnormal, clinically relevant laboratory values not related to RA
* Participation in another clinical trial during this study or during the previous month
* Previous participation in this trial (i.e. having been allocated a randomized treatment number)
* Patient unable to comply with the protocol
* Patient with known drug abuse
* Patient with known alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2000-01; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Mac-1 expression | Pre-dose, up to day 14 after start of treatment
Plasma concentrations of BIIL 284 BS, BIIL 260 BS, BIIL 315 ZW and BIIL 304 ZW | Pre-dose, up to day 14 after start of treatment
Maximum concentration of the analyte in plasma (Cmax) | Pre-dose, up to day 14 after start of treatment
Trough concentration of the analyte in plasma shortly before drug administration in a steady state dosing interval (Cpre,ss) | Pre-dose, up to day 14 after start of treatment
Time to reach the maximum concentration of the analyte in plasma (tmax) | Pre-dose, up to day 14 after start of treatment
Area under the concentration-time curve of the analyte in plasma (AUC) | Pre-dose, up to day 14 after start of treatment
Number of patients with adverse events | Up to 4 weeks
Global assessment of tolerability by the patient on a 4-point scale | Up to 14 days after start of treatment
Global assessment of tolerability by investigator on a 4-point scale | Up to 14 days after start of treatment

SECONDARY OUTCOMES:
Changes from baseline in tender joint count (TJC) | Pre-dose, up to day 14 after start of treatment
  Bilateral assessment of twenty-eight joints by e.g., pressure, joint manipulation etc.
Changes from baseline in swollen joint count (SJC) | Pre-dose, up to day 14 after start of treatment
  Twenty-eight joints were bilaterally assessed whether they are swollen or not
Changes from baseline in patient's current pain level assessment by visual analogue scale (VAS) | Pre-dose, up to day 14 after start of treatment
Changes from baseline in patient's global assessment of disease activity by VAS | Pre-dose, up to day 14 after start of treatment
Global assessment of disease activity by investigator on a 5-point scale | Up to 14 days after start of treatment
Changes from baseline for patient's assessment of physical function | Pre-dose, up to day 14 after start of treatment
  Functional disability was measured using the disability section of the Health Assessment Questionnaire (HAQ)
Changes from baseline in erythrocyte sedimentation rate (ESR) | Pre-dose, up to day 14 after start of treatment
Changes from baseline in C-reactive protein (CRP) | Pre-dose, up to day 14 after start of treatment
Changes from baseline in american college of rheumatology (ACR) 20 score | Pre-dose, up to day 14 after start of treatment
Changes from baseline in disease activity score (DAS) | Pre-dose, up to day 14 after start of treatment
Global efficacy assessment by the patient on a 4-point scale | Up to 14 days after start of treatment
Number of withdrawals due to adverse events | Up to 4 weeks
Number of patients with clinically significant findings in laboratory adverse events | Up to 4 weeks
Number of patients with clinically significant findings in vital signs (blood pressure, pulse rate) | Up to 4 weeks